CLINICAL TRIAL: NCT00555399
Title: Phase I / II Adaptive Randomized Trial of Vorinostat, Isotretinoin and Temozolomide in Adults With Recurrent Glioblastoma Multiforme
Brief Title: Vorinostat, Isotretinoin and Temozolomide in Adults With Recurrent Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No Sponsor funding for continuation of trial
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0709; NCI-2010-00782 (Registry Identifier: NCI CTRP); 4808704; BTTC09-02 (Other: Brain Tumor Trials Collaborative (BTTC))
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme; Anaplastic Glioma
Keywords: Glioblastoma Multiforme; Anaplastic Glioma; Vorinostat; Suberoylanilide Hydroxamic Acid; SAHA; MSK-390; Zolinza; Isotretinoin; Accutane; 13-cis-Retinoic Acid; Carboplatin; Paraplatin; CBT; Temozolomide; Temodar
MeSH Terms: conditions — Glioblastoma | interventions — Vorinostat; Isotretinoin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ph I: Arm 1 (Experimental): Vorinostat plus isotretinoin
  Interventions: Drug: Vorinostat; Drug: Isotretinoin
- Ph I: Arm 2 (Experimental): Temozolomide plus isotretinoin
  Interventions: Drug: Isotretinoin; Drug: Temozolomide
- Ph I: Arm 3 (Experimental): Vorinostat plus isotretinoin plus temozolomide
  Interventions: Drug: Vorinostat; Drug: Isotretinoin; Drug: Temozolomide
- Ph II: Arm 1 (No Intervention): Non-Surgical
- Ph II: Arm 2 (Other): Surgical Arm
  Interventions: Procedure: Surgical Resection

INTERVENTIONS:
Drug: Vorinostat — Phase I/Arm 1: Level 0 = 300 mg PO x 14 days; Level I = 400 mg PO x 14 days; Level II = 500 mg PO x 14 days.
  Phase I/Arm 3: Level -II = 300 mg PO x 14 days; Level -I = 400 mg PO x 14 days; Level 0 = 400 mg PO x 14 days; Level I = 500 mg PO x 14 days.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
  Arms: Ph I: Arm 1; Ph I: Arm 3
Drug: Isotretinoin — Phase I/Arm 1: Level 0 = 100 mg/m^2/day PO x 21 days; Level I = 100 mg/m^2/day PO x 21 days; Level II = 100 mg/m^2/day PO x 21 days.
  Phase I/Arm 2: Level 0 = 100 mg/m^2/day PO x 21 days; Level I = 100 mg/m^2/day PO x 21 days; Level II = 100 mg/m^2/day PO x 21 days.
  Phase I/Arm 3: Level -II = 100 mg/m^2/day PO x 21 days; Level -I = 100 mg/m^2/day PO x 21 days; Level 0 = 100 mg/m^2/day PO x 21 days; Level I = 100 mg/m^2/day PO x 21 days; Level II = 100 mg/m^2/day PO x 21 days.
  Other Names: cRA; Accutane; 13-cis-Retinoic Acid
  Arms: Ph I: Arm 1; Ph I: Arm 2; Ph I: Arm 3
Procedure: Surgical Resection — Surgical Resection for recurrent Glioblastoma Multiforme
  Arms: Ph II: Arm 2
Drug: Temozolomide — Phase I/Arm 2: All Levels = 150 mg/m2/day PO X 14 days.
  Phase I/Arm 3: Level 0 = 150 mg/m2/day PO X 14 days; Level I = 150 mg/m2/day PO X 14 days; Level -I = 125 mg/m2/day PO X 14 days; Level -II = 125 mg/m2/day PO X 14 days; Level -III = 100 mg/m2/day PO X 14 days.
  Other Names: Temodar
  Arms: Ph I: Arm 2; Ph I: Arm 3

SUMMARY:
The goal of this clinical research study is to learn if vorinostat when given with isotretinoin and temozolomide can help to control glioblastoma or gliosarcoma. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 3 groups. If you are on of the first 30 participants in the study, you will be randomly assigned to a group. If you are enrolled after the first 30 participants, you will be more likely to be enrolled in the group that is showing better results.

* If you are in Group 1, you will take vorinostat and isotretinoin.
* If you are in Group 2, you will take isotretinoin and temozolomide.
* If you are in Group 3, you will take vorinostat, isotretinoin and temozolomide.

Study Drug Administration:

Each study cycle is 28 days.

You will take vorinostat by mouth once a day during Days 1-7 and Days 15-21 of each cycle. You should take vorinostat by mouth in the morning, at about the same time each day. Vorinostat capsules should be swallowed whole and should not be opened. If a capsule is damaged or broken, spills of powder from vorinostat capsules should be cleaned up carefully. If you come in contact with the powder, you should wash your hands thoroughly. If the spill is on a surface, the area must be washed at least 3 times with rubbing alcohol, followed by water. Vorinostat capsules should be stored at room temperature (59°-86°F [15°-30°C]) in a dry area. You should take vorinostat with food, but not a high fat meal.

You will also take isotretinoin by mouth 2 times a day on Days 1-21 of each cycle.

You will take temozolomide by mouth once a day on Days 1-7 and Days 15-21 of each cycle. You should take temozolomide by mouth at bedtime, at about the same time each day. You should swallow the temozolomide capsules whole, one right after the other, without chewing them. They should be taken on an empty stomach (at least 2 hours after eating) with 1 cup (about 8 ounces) of water.

If you vomit while taking vorinostat, isotretinoin and/or temozolomide, you should not "make up" the dose. You should wait until the next scheduled dose.

Study Visits:

At Week 2 of every cycle:

° Blood (about 1 teaspoons) will be drawn for routine tests.

At Week 4 of Cycles 1:

* Blood (about 2 teaspoons) will be drawn for routine tests and to check how well your blood clots,.
* If you are able to become pregnant, you will have a blood (about 1/2 teaspoon) pregnancy test.

At Week 4 of Cycle 2 and then every other cycle after that (Cycles 4, 6, 8, and so on):

* You will have a physical exam, including a neurological exam.
* Blood (about 2 teaspoons) will be collected for routine tests. This routine blood draw will also include a pregnancy test if you can become pregnant.
* Blood (about 2 teaspoons) will be drawn to check how well your blood clots, your pancreas function and the amount of fats in your blood.
* You will have a brain MRI scan to check the status of the disease.

At any time during the study, extra tests may be performed if the doctor thinks they are needed for your safety. The study doctor will tell you more about any extra tests.

Length of Study:

You may take the study drug(s) for up to 1 year. You may continue to receive the study drug(s) beyond 1 year if your doctor decides that it is in your best interest. You will be taken off study early if the disease gets worse or you have intolerable side effects.

Long-Term Follow-Up:

After your last dose of the study drug, every 2 months after that, you may be called and asked how you are feeling. This phone call should take about 5-10 minutes.

If you stop the study drugs because of intolerable side effects, you will visit the clinic every 2 months, unless the disease gets worse. At these visits, You will have a physical exam, including a neurological exam.

* Blood (about 2 teaspoons) will be collected for routine tests. This routine blood draw will also include a pregnancy test if you can become pregnant.
* Blood (about 2 teaspoons) will be drawn to check how well your blood clots, your pancreas function and the amount of fats in your blood.
* You will have a brain MRI scan to check the status of the disease.

This is an investigational study. Isotretinoin, temozolomide, and vorinostat are FDA approved drugs and commercially available. The use of these drugs in this combination is investigational.

Up to 135 patients will take part in this study. Up to 30 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven supratentorial WHO grade IV glioma (glioblastoma or gliosarcoma) will be eligible for the study.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan and should have failed radiation therapy. The scan done prior to study entry documenting progression will be reviewed by the treating physician to document changes in tumor dimension to confirm recurrence. Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis.
3. (2. continued) Patients with prior therapy that included interstitial brachytherapy, Gliadel wafers or stereotactic radiosurgical procedures must have confirmation of true progressive disease rather than radiation necrosis. Such confirmation may be using advanced imaging studies (e.g. PET scans, diffusion-perfusion MRI, SPECT etc) or if available, surgical sampling and histological confirmation (surgery is not required).
4. Patients may have had up to 2 prior relapses.
5. All patients must sign an IRB approved informed consent indicating their awareness of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
6. The baseline on-study MRI should be performed within 14 days (+ 3 working days) prior to registration and on a steroid dosage that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and the initiation of therapy (or at that time), a new baseline MRI is required. The same type of scan, i.e., MRI, must be used throughout the period of protocol treatment for tumor measurement.
7. Patients who have undergone recent resection of recurrent or progressive tumor will be eligible as long as they have recovered from the effects of surgery. Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual measurable disease post-operatively, a MRI should be done no later than 96 hours in the immediate post-operative period or 4-6 weeks post-operatively.
8. Patients must be 18 years old or older.
9. Patients must have a Karnofsky performance status equal or greater than 60.
10. Patients must have recovered from the toxic effects of prior therapy to < grade 2 non hematological or grade 2 or lesser hematological toxicity per CTC ver 4 (except deep vein thrombosis): 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count). Patients who receive anticancer agents for non-therapeutic purposes unrelated to this study
11. (10. continued) (such as presurgically for obtaining pharmacology data for the agent) will be eligible to enter the study provided they have recovered from the toxic effects of the agent if any. Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
12. Patients must have adequate bone marrow function (ANC = or > 1,500/mm^3 and platelet count of = or > 100,000/mm^3), adequate liver function (SGPT = or < 3 times upper limit of normal and alkaline phosphatase = or < 2 times upper limit of normal, bilirubin = or <1.5 mg/dl), adequate renal function (BUN and creatinine = or <1.5 times upper limit of normal) and normal serum amylase and lipase prior to starting therapy. Elevated cholesterol and triglycerides are not a contraindication to study enrollment, but should be managed as clinically appropriate by the treating physician.
13. Patients must be willing and able to comply with the FDA mandated iPLEDGE program for treatment with isotretinoin (cRA). Patients must sign specific informed consents for treatment with cRA, as mandated by iPLEDGE guidelines. Women of childbearing potential must not be pregnant, must not be breast-feeding and must practice adequate contraception during and one month after participation in the study. Male and Female patients on treatment with vorinostat must agree to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication.
14. Prior treatment with dose dense regimens of temozolomide is not allowed (e.g, 7 days on/7 days off, 21 day/28 day and daily low dose continuous dosing). However, prior treatment with standard day 1-5 dosing in the adjuvant setting and low dose daily dosing as part of chemoradiation therapy are allowed
15. Prior treatment with isotretinoin is allowed because the trial is based on the hypothesis that HDAC inhibition will potentially overcome resistance to retinoids.

Exclusion Criteria:

1. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix or bladder), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
2. Patients must not have: a) active infection; b) disease that will obscure toxicity or dangerously alter drug metabolism, especially liver disease; c) serious intercurrent medical illness; d) prior treatment with HDAC inhibitors. However, patients who have received anticancer agents for non-therapeutic purposes (for eg., as part of a pharmacology study without therapeutic intent) will remain eligible for enrollment into the study.
3. Prior treatment with bevacizumab is not allowed.
4. Patients receiving valproic acid (VPA), an anticonvulsant drug with HDAC inhibitor properties, will be excluded, unless they are switched to an alternative agent prior to treatment initiation. No wash out period is required.
5. Patients on previous treatment with carboplatin.
6. Patients with a known allergy to any component of vorinostat, or a known allergy to temozolomide and/or isotretinoin.
7. Patient must be able to tolerate the procedures required in this study including periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study. Inability to comply with protocol or study procedures (for example, an inability to swallow tablets) will be an exclusion criterion.
8. Patients receiving treatment with other antiepileptic medications will not be excluded. Vorinostat is not metabolized by cytochrome P450 3A4 (CYP 3A4). However, vorinostat may potentially suppress CYP 3A4 activity. Therefore, patients should preferably be treated with non-enzyme inducing anti-epileptic medications to avoid any potential interactions with vorinostat.
9. (8. continued) However, the use of non-enzyme inducing anti-epileptic medications is not mandatory. If enzyme-inducing antiepileptic drugs are used, monitoring of drug levels should be considered, as considered clinically appropriate by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-11-28 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Penas-Prado, MD, Principal Investigator — M.D. Anderson Cancer Center; Vinay Puduvalli, MD, Study Chair — Brain Tumor Trials Collaborative (BTTC), and Ohio State University
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 participants were enrolled .
Groups:
- Arm 1 Cohort 1: Cohort1= VOR 300mg/day D1-14, Each Cohort also had set cRA 100mg/m2/day D1-2
- Arm 1 Cohort 2: Cohort 2=VOR 400 mg/day D1-14, Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 1 Cohort 3; Arm 2 Cohort 1: Cohort 3=VOR 500mg/day D1-14; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 2 Cohort 2: CBT: Cohort2= AUC5 D1; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 2 Cohort 3: CBT: Cohort3= AUC6 D1; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 3A Cohort 1: Cohort1=Vor 400 mg/day x14 days; CBT AUC 6; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3A Cohort 2: Cohort2=Vor 400 mg; /day x14 days; CBT AUC 5; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3A Cohort 3: Cohort3=Vor 300mg/day x14 days; CBT AUC5 Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3A Cohort 4: Cohort4=Vor 300 mg/day x14 days; CBT AUC 4; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3B Cohort 1: Cohort 1=Vor 400 mg/day, D 1-7 & 15-21; Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21"
- Arm 3B Cohort 2: Cohort 2=Vor 500 mg/day, D 1-7 & 15-21 Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21
Period: Overall Study
Arm/Group | Arm 1 Cohort 1 | Arm 1 Cohort 2 | Arm 1 Cohort 3 | Arm 2 Cohort 1 | Arm 2 Cohort 2 | Arm 2 Cohort 3 | Arm 3A Cohort 1 | Arm 3A Cohort 2 | Arm 3A Cohort 3 | Arm 3A Cohort 4 | Arm 3B Cohort 1 | Arm 3B Cohort 2
Started | 3 | 3 | 8 | 6 | 3 | 3 | 5 | 6 | 5 | 3 | 3 | 7
Completed | 3 | 3 | 6 | 6 | 3 | 3 | 5 | 6 | 5 | 3 | 3 | 6
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient decided not to proceed with treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data provided for the demographics of participants enrolled into each arm is not related to the treatment cohorts but to the combination of agents used.
Groups:
- Arm 1 Cohort 1: Cohort1= VOR 300mg/day D1-14, Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 2 Cohort 1: CBT: Cohort1= AUC4 D1; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 3B Cohort 1: Cohort 1=Vor 400 mg/day, D 1-7 & 15-21; Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21
- Total: Total of all reporting groups
Arm/Group | Arm 1 Cohort 1 | Arm 1 Cohort 2 | Arm 1 Cohort 3 | Arm 2 Cohort 1 | Arm 2 Cohort 2 | Arm 2 Cohort 3 | Arm 3A Cohort 1 | Arm 3A Cohort 2 | Arm 3A Cohort 3 | Arm 3A Cohort 4 | Arm 3B Cohort 1 | Arm 3B Cohort 2 | Total
Number analyzed (Participants) | 3 | 3 | 8 | 6 | 3 | 3 | 5 | 6 | 5 | 3 | 3 | 7 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 6 | 3 | 3 | 4 | 4 | 5 | 3 | 2 | 5 | 46
  >=65 years | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 4 | 1 | 2 | 2 | 3 | 3 | 1 | 2 | 1 | 23
  Male | 1 | 3 | 6 | 2 | 2 | 1 | 3 | 3 | 2 | 2 | 1 | 6 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 2 | 2 | 6 | 5 | 1 | 3 | 4 | 5 | 2 | 3 | 3 | 7 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 8 | 6 | 3 | 3 | 5 | 6 | 5 | 3 | 3 | 7 | 55

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: To determine the maximum tolerated dose (MTD) of vorinostat + isotretinoin (cRA), carboplatin (CBT) + cRA, and vorinostat + cRA + CBT combinations in adult patients with recurrent glioblastoma multiforme (GBM) and anaplastic gliomas. The units of measurement for the drug dose were either mg/day [VOR and cRA] or AUC [CBT]. In the outcome measure data table below we have provided the cohort number for each arm at which MTD was declared.
Time Frame: 62 months
Population: 52 out of 55 enrolled participants were evaluable. Two patients withdrew consents, and one patient chose not to proceed with treatment.
Measure: Number; unit: cohort number
Groups:
- Arm 1 (MTD Cohort Number): Cohort1= VOR 300mg/day D1-14, Cohort 2=VOR 400 mg/day D1-14, Cohort 3=VOR 500mg/day D1-14; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 2 (MTD Cohort Number): CBT: Cohort1= AUC4 D1; Cohort2= AUC5 D1; Cohort3= AUC6 D1; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 3A (MTD Cohort Number): Cohort1=Vor 400 mg/day x14 days; CBT AUC 6; Cohort2=Vor 400 mg; /day x14 days; CBT AUC 5; Cohort3=Vor 300mg/day x14 days; CBT AUC5 Cohort4=Vor 300 mg/day x14 days; CBT AUC 4; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3B (MTD Cohort Number): Cohort 1=Vor 400 mg/day, D 1-7 & 15-21; Cohort 2=Vor 500 mg/day, D 1-7 & 15-21 Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21"
Arm/Group | Arm 1 (MTD Cohort Number) | Arm 2 (MTD Cohort Number) | Arm 3A (MTD Cohort Number) | Arm 3B (MTD Cohort Number)
Number analyzed (Participants) | 12 | 12 | 19 | 9
cohort number | 2 | 2 | 4 | 2

2. Primary Outcome: Phase II: To Determine the Efficacy of Vorinostat + cRA, Versus CBT + cRA, Versus Vorinostat + cRA + CBT in Patients With Recurrent Glioblastoma Multiforme as Determined by Time to Progression (TTP) Using an Adaptive Randomization Phase II Trial Design.
Description: Phase II of the trial has never opened d/t Sponsor's withdrawal of the funding
Time Frame: two patients withdrew consents and one pt chose not to proceed with treatment
Population: two patients withdrew consents and one pt chose not to proceed with treatment
Groups:
- Arm 1 (CRA+VOR 300mg or VOR 400 mg or VOR 500mg): Cohort1= VOR 300mg/day D1-14, Cohort 2=VOR 400 mg/day D1-14, Cohort 3=VOR 500mg/day D1-14; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 2 (CRA+CBT AUC4 or AUC5 or AUC6): CBT: Cohort1= AUC4 D1; Cohort2= AUC5 D1; Cohort3= AUC6 D1; Each Cohort also had set cRA 100mg/m2/day D1-21
- Arm 3A(CRA+Vor400 mg+CBT AUC6 or Vor400 mg+CBT AUC 5 or Vor 300 mg+CBT AUC 5 or Vor300 mg+CBT AUC 5): Cohort1=Vor 400 mg/day x14 days; CBT AUC 6; Cohort2=Vor 400 mg; /day x14 days; CBT AUC 5; Cohort3=Vor 300mg/day x14 days; CBT AUC5 Cohort4=Vor 300 mg/day x14 days; CBT AUC 4; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3B (CRA+TMZ+Vor 400 mg or Vor 500): Cohort 1=Vor 400 mg/day, D 1-7 & 15-21; Cohort 2=Vor 500 mg/day, D 1-7 & 15-21 Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21"
Arm/Group | Arm 1 (CRA+VOR 300mg or VOR 400 mg or VOR 500mg) | Arm 2 (CRA+CBT AUC4 or AUC5 or AUC6) | Arm 3A(CRA+Vor400 mg+CBT AUC6 or Vor400 mg+CBT AUC 5 or Vor 300 mg+CBT AUC 5 or Vor300 mg+CBT AUC 5) | Arm 3B (CRA+TMZ+Vor 400 mg or Vor 500)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 65 months
Groups:
- Arm 3A Cohort 4: Cohort4=Vor 300 mg/day x14 days; CBTP AUC 4; Each Cohort also had set cRA 100 mg/m2/day x 21 days
- Arm 3B Cohort 2: Cohort 2=Vor 500 mg/day, D 1-7 & 15-21 Each Cohort also had set cRA 100 mg/m2/day, D 1-21 & TMZ 150 mg/m2/day, D 1-7 &15-21"
Arm/Group | Arm 1 Cohort 1 | Arm 1 Cohort 2 | Arm 1 Cohort 3 | Arm 2 Cohort 1 | Arm 2 Cohort 2 | Arm 2 Cohort 3 | Arm 3A Cohort 1 | Arm 3A Cohort 2 | Arm 3A Cohort 3 | Arm 3A Cohort 4 | Arm 3B Cohort 1 | Arm 3B Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/8 | 0/6 | 0/3 | 0/3 | 0/5 | 1/6 | 0/5 | 0/3 | 0/3 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/8 | 0/6 | 0/3 | 0/3 | 0/5 | 1/6 | 0/5 | 0/3 | 0/3 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 6/6 | 3/3 | 3/3 | 5/5 | 6/6 | 5/5 | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Cohort 1 (N=3) | Arm 1 Cohort 2 (N=3) | Arm 1 Cohort 3 (N=8) | Arm 2 Cohort 1 (N=6) | Arm 2 Cohort 2 (N=3) | Arm 2 Cohort 3 (N=3) | Arm 3A Cohort 1 (N=5) | Arm 3A Cohort 2 (N=6) | Arm 3A Cohort 3 (N=5) | Arm 3A Cohort 4 (N=3) | Arm 3B Cohort 1 (N=3) | Arm 3B Cohort 2 (N=7)
Pulmonary Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Cohort 1 (N=3) | Arm 1 Cohort 2 (N=3) | Arm 1 Cohort 3 (N=8) | Arm 2 Cohort 1 (N=6) | Arm 2 Cohort 2 (N=3) | Arm 2 Cohort 3 (N=3) | Arm 3A Cohort 1 (N=5) | Arm 3A Cohort 2 (N=6) | Arm 3A Cohort 3 (N=5) | Arm 3A Cohort 4 (N=3) | Arm 3B Cohort 1 (N=3) | Arm 3B Cohort 2 (N=7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 | 3 | 6 | 2 | 3 | 3 | 3 | 5 | 4 | 2 | 3 | 6
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 2 | 4 | 1 | 1 | 1
Platelets count decreased (Blood and lymphatic system disorders) | 1 | 1 | 5 | 3 | 2 | 2 | 4 | 4 | 3 | 2 | 3 | 5
Cholesterol Elevated (Cardiac disorders) | 2 | 2 | 5 | 6 | 1 | 2 | 5 | 6 | 4 | 3 | 2 | 3
Dyspnea (Cardiac disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 3
Alopecia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 4 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 3 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 4 | 1 | 2 | 2 | 1 | 5 | 1 | 2 | 5
Vomitting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1
ALT elevated (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1
AST elevated (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Fatigue (Nervous system disorders) | 3 | 2 | 4 | 4 | 3 | 3 | 5 | 1 | 3 | 1 | 2 | 6
Insomnia (Nervous system disorders) | 2 | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 5 | 2 | 1 | 3 | 0 | 4 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-03-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT00555399/Prot_SAP_000.pdf